CLINICAL TRIAL: NCT07061574
Title: A Randomized Phase 1/2 Trial of Low Dose Anti-thymocyte Globulin (ATG) With Subsequent Adalimumab or Verapamil in New Onset Type 1 Diabetes
Acronym: WAVE T1D
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: Jaeb Center for Health Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 24745
Record Dates: First submitted 2025-07-02; First posted 2025-07-11 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Type 1 Diabetes; New Onset
Keywords: ATG, Verapamil, Adalimumab
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Antilymphocyte Serum; thymoglobulin; Adalimumab

STUDY DESIGN:
Intervention Model Description: Multi-center, randomized, double blind, placebo-controlled phase 1/2 clinical trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants will be randomized 2:2:1:1 using blocked randomization to ATG + Adalimumab, ATG + Verapamil, ATG + injectable placebo, ATG + oral placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- ATG + Placebo (Placebo Comparator): ATG (brand name Thymoglobulin) a polyclonal T cell antibody preparation. It will be given at low doses (0.5 mg/kg Day 1 then 2 mg/kg Day 2). This group will receive Verapamil (Oral) placebo or Adalimumab (injectable) placebo.
  Interventions: Drug: Anti-thymocyte globulin (ATG)
- ATG + Verapamil (Experimental): Low dose ATG (0.5 mg/kg Day 1 then 2 mg/kg Day 2). From the 6-week visit until the 156-week visit, daily oral administration at 60, 120, 240 or 360 mg based on weight and ECG findings.
  Interventions: Drug: verapamil extended-release capsule
- ATG + Adalimumab (Experimental): Low dose ATG (0.5 mg/kg Day 1 then 2 mg/kg Day 2). From the 6-week visit until the 156-week visit, Participants will receive a 40 mg dose injection every other week.
  Interventions: Drug: Adalimumab

INTERVENTIONS:
Drug: Anti-thymocyte globulin (ATG) — ATG (brand name Thymoglobulin) a polyclonal T cell antibody preparation. The first dose (0.5 mg/kg) will be infused on day 0, during a period of 6 hours. The second dose (2 mg/kg) will be given on day 1, over a period of 4 to 6 hours.
  Other Names: Thymoglobulin
  Arms: ATG + Placebo
Drug: verapamil extended-release capsule — Daily oral (pill) administration at 60, 120, 240 or 360 mg based on weight and ECG findings.
  Arms: ATG + Verapamil
Drug: Adalimumab — 40 mg administered subcutaneously every other week beginning 6 weeks after the last dose of ATG until the 156-week visit.
  Other Names: Simlandi
  Arms: ATG + Adalimumab

SUMMARY:
This multi-center randomized controlled trial will assess the safety and efficacy of ATG followed by either adalimumab or verapamil in preserving insulin secretion 2 years from randomization in persons aged 9 to <21 with recent-onset stage 3 T1D.

DETAILED DESCRIPTION:
The primary objective of this study is to assess the safety and efficacy of ATG followed by either adalimumab or verapamil in preserving insulin secretion 2 years from randomization in persons with T1D. The secondary objectives are to assess metabolic and safety endpoints at 2 years and at timepoints between baseline and two years.

ELIGIBILITY:
Key Inclusion Criteria:

Recent-onset stage 3 T1D diagnosed by standard ADA criteria, with the ability to be randomized within 6 months from the date of T1D diagnosis and within 37 days of Screening Visit.

* At least one positive T1D auto-antibody.
* If clearly positive (≥20% above local lab's ULN) at screening, repeat antibody testing for central lab is not required.
* Insulin auto-antibodies are only considered if exogenous insulin use is <10 days when blood is drawn.
* Must have stimulated C-peptide levels ≥0.2 pmol/mL measured during MMTT conducted prior to randomization.
* Age 9 to <21 years at the time of randomization.
* Body weight >30kg.
* BMI <95th percentile for age and gender.
* Willing to comply with intensive diabetes management.
* Female participants with childbearing potential are not currently pregnant, are willing to avoid pregnancy and breastfeeding, and to undergo pregnancy testing prior to MMTTs for the duration of the study.
* Women of childbearing potential (WOCBP) must use an acceptable form of birth control. Acceptable forms include oral/injection contraceptives, transdermal contraceptives, diaphragm, intrauterine devices, condoms with spermicide, documented surgical sterilization of either the participant or their partner or abstinence.
* Male participants with potential to father children must be willing to use abstinence or adequate contraceptive methods for the duration of the study.
* Males must agree to be sexually abstinent or use a condom and agree not to donate sperm for the treatment period and for a minimum of 1 spermatogenesis cycle (90 days after last dose of study drug) after last treatment.
* Willing to provide informed consent and child assent as applicable.
* Sufficient cognitive ability, per investigator judgment, to provide informed consent for study participation on an IRB approved consent form.
* Able to read and understand English or Spanish (both participant and legally authorized representative, if applicable).
* Must be fully vaccinated for age.
* Must have been vaccinated for flu (if currently in flu season).
* Must be willing to not receive live vaccines throughout the treatment period.
* Must be willing to not use any non-insulin glucose-lowering agents such as GLP-1 agonists (including for weight loss indication), symlin, DPP-4 inhibitors, SGLT-2 inhibitors, biguanides, sulfonylureas) for the duration of study treatment. Participants are required to go off these drugs at least 30 days prior to screening.

Key Exclusion Criteria:

* Prior treatment with ATG or known allergy to ATG or rabbit-derived products.
* Local lab draw at screening:
* Immunodeficient or have clinically significant chronic lymphopenia: Leukopenia (<3,000 leukocytes /μL), neutropenia (<1,500 neutrophils/μL), lymphopenia (<800 lymphocytes/μL).
* Thrombocytopenia (<100,000 platelets/μL) or anemia (hemoglobin < 10g/dL).
* Leukocytosis (>14,000/mL)
* Infections:
* Ongoing infection or had recently had a major infection requiring hospitalization or intravenous antibiotics.within 30 days prior to randomization.
* Have active signs or symptoms of acute infection at the time of randomization.
* Have evidence of prior or current tuberculosis infection as assessed interferon gamma release assay (QuantiFERON), or a positive test for latent tuberculosis.
* Have evidence of current or past HIV or Hepatitis B or current Hepatitis C infection.
* History of serious bacterial, viral, fungal, or other opportunistic infections.
* Have active signs or symptoms of CMV or EBV compatible illness lasting more than 7 days within 30 days of randomization.
* Have positive CMV and/or EBV PCR test within 30 days prior to randomization.
* Have positive COVID-19 self-antigen test within 3 days of randomization.
* History of underlying cardiac disease (ex. left ventricular dysfunction, hypertrophic cardiomyopathy), certain arrhythmias (e.g. AV block, accessory pathway such as Wolff- Parkinson-White or Lown-Ganong-Levine syndromes) or abnormal ECG (unless cleared by cardiology).
* Blood pressure (either systolic or diastolic) <5th percentile for age, gender, and height on two out of three measurements.
* Pulse <2nd percentile for age and gender on two out of three measurements.
* History of vasovagal syncopal episodes related to hypotension.
* History of malignancies other than of skin.
* Use of medications likely to interfere with study results:
* Any immunomodulators, including systemic steroids or participation in prior research study in which a potential participant received an immunomodulatory agent (may participate if received placebo only).
* Current or previous use of Teplizumab.
* Ongoing use of medications known to influence glycemia or glucose tolerance. Only topical steroids are allowed.
* Need to use of any of the following medications during the study: beta blocker, seizure medication (carbamazepine, phenobarbital, phenytoin), other antihypertensive medications, HMG-CoA reductase inhibitors, lithium, theophylline, clonidine.
* Receipt of live vaccine (e.g., varicella, measles, mumps, rubella, cold-attenuated intranasal influenza vaccine, bacillus Calmette-Guerin, and smallpox) within the 90 days before randomization.
* Any known hypersensitivity reaction to any of the study medications or their components.
* Unable to swallow pills (tested with an inert imitation tablet in clinic at screening).
* History of significant allergy (e.g., anaphylaxis) to milk or soy proteins in the Boost drink required for study MMTT testing.
* Current use of hydroxyurea or unable to avoid hydroxyurea use during the study (interferes with accuracy of Dexcom sensor).
* Established history of allergy or severe reaction to adhesive or tape that must be used in the study.
* Participation in another treatment research study that involves diabetes care or immune modulation, unless the participant is able to confirm that they were in the placebo arm.
* Presence of a medical condition or use of a medication that, in the judgment of the investigator, clinical protocol chair, or medical monitor, could compromise the results of the study or the safety of the participant. Conditions to be considered by the investigator may include the following:
* Alcohol or drug abuse
* Untreated or inadequately treated mental illness
* Liver disease or LFTs >2x ULN.
* Renal disease or creatinine greater than 1.5x ULN.
* Other autoimmune diseases except for stable and treated hypothyroidism
* Graves' disease, or celiac disease (e.g., symptom-free on a gluten free diet).
* Nervous system disorder including but not limited to Guillain-Barre
* Syndrome, multiple sclerosis, progressive multifocal leukoencephalopathy.
* History of multiple abdominal surgeries and/or at increased risk for bowel obstruction.
* Any clinical or laboratory conditions that the investigator feels would interfere with the study or participant safety (e.g., increased risk to pre-existing disease).

Any lab abnormality believed to be transient may be repeated at the discretion of the site PI. If repeat value does not preclude participation, and potential participant would otherwise qualify for the study, then may proceed with enrollment per investigator discretion.

-

Ages: 9 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2030-04-15 (Estimated); Study Completion 2031-04-15 (Estimated)

PRIMARY OUTCOMES:
Stimulated C-peptide AUC | Week 104
  The primary outcome is the C-peptide in response to a 2-hour MMTT at week 104. This is measured as the area under the stimulated C-peptide curve (AUC). AUC is computed using a trapezoidal rule, which is a weighted sum of the C-peptide values over 120 minutes.

SECONDARY OUTCOMES:
Severe Adverse Events | week13, week 26, week 52, week 78, and week 104
  Prevalence of SAE of grade 3 or above, that may be attributable to study medications at all follow-up time points.
Adverse Events | Week 104
  Number and severity of AEs.
Severe Hypoglycemia | Week 104
  Rate of severe hypoglycemia, defined as an event requiring assistance of another person due to altered consciousness and another person to actively administer carbohydrate, glucagon, or other resuscitative actions.
Diabetic ketoacidosis (DKA) | Week 104
  Number of DKA events (rate assessed if sufficient events)
Number of Participants with CD4 count <500 mm3 | Week 104
  Frequency of CD4 count <500 mm3
Number of Participants with Total Lymphocyte count <800/mm3 | Week 104
  Frequency of Total Lymphocyte count <800/mm3

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Pugliese, MD, Study Chair — City of Hope Medical Center
Locations (11):
- United States (11):
  - UCSF, San Francisco, California
  - Barbara Davis Center for Diabetes University of Colorado Anschutz, Aurora, Colorado
  - Yale University, New Haven, Connecticut
  - University of Florida, Gainesville, Florida
  - University of Miami, Miami, Florida
  - Indiana University, Indianapolis, Indiana
  - University of Minnesota, Minneapolis, Minnesota
  - University of Buffalo, Buffalo, New York
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided
Undecided yet